CLINICAL TRIAL: NCT03987659
Title: A Randomised Controlled Pilot Study to Determine the Effect of Irrigation Techniques Used to Enhance the Release of Endogenous Signalling Molecules From Dentine Matrix to Treat Apical Periodontitis
Brief Title: Therapeutic Irrigation Procedures to Treat Apical Periodontitis
Acronym: TIPTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG_19-062
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root Canal Treatment without dECMs release (Active Comparator): Two visit non-surgical root canal therapy with conventional irrigation protocols
  Interventions: Procedure: Conventional Irrigation protocols
- Root Canal Treatment with dECMs release (Experimental): Two visit non-surgical root canal treatment with irrigation protocols that optimise release of soluble dentine extracellular matrix components (dEMCs)
  Interventions: Procedure: Irrigation protocols that promote release of dECMs

INTERVENTIONS:
Procedure: Irrigation protocols that promote release of dECMs — Irrigation protocols that promote release of dECMs
  Arms: Root Canal Treatment with dECMs release
Procedure: Conventional Irrigation protocols — Conventional Irrigation protocols
  Arms: Root Canal Treatment without dECMs release

SUMMARY:
Apical periodontitis is a dental infection which develops around the root of a tooth and affects ~4-6% of the UK population. Current treatment strategies focus solely on removing bacteria from within the root canal space during Non-Surgical Root Canal Treatment (NSRCT). Despite radical improvements in techniques available to disinfect canals, over the last 2-3 decades there has been no proportionate improvement in success rates, with ~20% of cases failing to demonstrate complete healing following NSRCT. Over time this has placed significant burden on public resources as evidenced by increased referrals to dental hospitals, extensive waiting lists and increased use of anti-microbials.

It has long been known numerous bioactive molecules (dentine extracellular matrix components [dECM]) exist within the structure of the dentine. In a laboratory setting, they have demonstrated significant antibacterial properties and the ability to induce the functional processes of dental tissue repair. Through a different irrigation procedure, this research group have optimised methods for releasing dECMs during NSRCT and hypothesise this intervention could potentially promote a reduction in inflammation, improve healing and lead to more favourable outcomes for patients suffering from apical periodontitis, a concept which has not yet been investigated. It is proposed that to test this hypothesis at the Birmingham Dental Hospital by comparing clinical/radiographic signs of periradicular healing, and the molecular inflammatory response, in patients undergoing standard NSRCT (control arm) to those who having NSRCT with an irrigant regime that promotes release of dEMCs (intervention arm).

Data generated from this randomised controlled pilot study will not only help to understand the process of healing following treatment of apical periodontitis at a molecular level, but also help to explore if there is therapeutic potential in enhancing dEMC release during NSRCT.

DETAILED DESCRIPTION:
- Introduction Apical periodontitis (AP) is an inflammatory condition of the periodontium that exists when there is a dynamic equilibrium between putative endodontic microorganisms and host defence mechanisms.

The ideal objective for treating this disease is to restore architecture and functions of the periradicular tissues that were lost to the immune response. Conventional therapies achieve these outcomes indirectly by reducing the microbial load within infected root canals to create a pro-healing environment. Whilst this approach may be enough to initiate periapical wound healing, which involves a highly co-ordinated sequence of haemostasis, inflammation, proliferation and remodelling, it offers no additional stimulus for biological regeneration thereafter. Unaided, these endogenous processes are often insufficient to achieve complete tissue regeneration and will instead be compensated by reparative scar tissue. Persistent periapical radiolucencies may therefore not only represent failure to eradicate intraradicular infection but also inadequate physiological regenerative processes, which could explain why larger lesions demonstrate higher treatment failure rates. It also suggests that to attain more predictable outcomes, it would be necessary to employ alternative strategies that simultaneously manage the microbial load and directly enhance intrinsic regenerative events within damaged periradicular tissues.

Stem cells are essential to wound healing processes as they possess high-proliferation rates, self-renewal capabilities and potential for multi-lineage differentiation. Embryonic stem cells are pluripotent as they can develop into stromal cells from any of the three germinal layers whereas multipotent postnatal stem cells are more restricted to organ-specific lineages. The latter are more amenable to clinical translation due to their autologous nature and presence within almost all adult tissues. A subset of multipotent progenitors derived from the mesoderm germ layer, called "mesenchymal stem cells" (MSC).has attracted particular interest within regenerative endodontics as they can give rise to several mineral producing mesoderm lineages, including bone. Moreover; whilst they are known to be harvested from bone-marrow, other reservoirs have been isolated from within the pulp and associated periodontal tissues of permanent and deciduous teeth. Named according to their tissue of origin, these "dental MSC" niches include "dental pulp stem cells" (DPSC), "stem cells from human exfoliated deciduous teeth" (SHED), "periodontal ligament stem cells" (PDLSC), "dental follicle precursor cells" (DFPC), "stem cells of the apical papilla" (SCAP), "gingival MSCs", "alveolar bone MSCs" and "tooth germ progenitor cells". When transplanted into in vivo human and animal models, these dental MSCs have demonstrated a potent capacity to regenerate pulp-like tissue in empty root canals, dentine-like tissues in endodontic perforation defects, and periodontal tissues in surgically created periodontal defects. Furthermore, the positive outcomes revealed from their applications to other non dento-alveolar tissues, including the treatment of autoimmune, cardiovascular, endocrine, hepatic, musculoskeletal, neurodegenerative, ophthalmic, dermatological and respiratory diseases, confirm their potential to be utilised as powerful therapeutic tools. Recent studies however have identified another clinically accessible dental MSC population directly within the inflamed periradicular tissues of infected mature permanent teeth. These periapical lesion-derived MSCs (PL-MSC) possess tremendous immunosuppressive and regenerative potential and could therefore provide exciting opportunities to develop therapies for AP that actively engage with the endogenous mechanisms of periradicular tissue regeneration.

The cellular events required for periradicular regeneration are co-ordinated by various growth factors, cytokines, chemokines and angiogenic and neurotrophic signalling molecules. Noteworthy examples include members of the Transforming Growth Factor-beta (TGF-β), Bone Morphogenetic Protein (BMP), Fibroblast Growth Factor (FGF) and Vascular Endothelial Growth Factor (VEGF) and Insulin Growth Factor (IGF) families amongst many. Whilst these polypeptides are endogenously secreted by host cells at the site of disease, they rapidly deplete due to their relatively short half-life within the extracellular environment. Fortunately, abundant reservoirs of these molecules are locally sequestered within the dentine's extracellular matrix. They are deposited by secreting odontoblasts during dentinogenesis and become fossilised during subsequent mineralisation. Thereafter, their bioactivity remains highly preserved through formation of proteoglycan bonds but these can be immediately reinstated upon release. This has previously been achieved on command through demineralising irrigants, pulp capping agents, epigenetic modifiers, and dental adhesives. The resulting extracts, formally termed "dentine extracellular matrix components" (dECM), have demonstrated a potent capacity to upregulate regenerative events within various odontogenic MSC niches. It is therefore plausible to expose PL-MSCs in situ to this cocktail of bioactive molecules to enhance local tissue healing. This approach could overcome current limitations associated with conventional treatments for AP and provide clinicians with unique capabilities to actively apply a biologically driven therapy to the diseased periradicular tissues.

- Research Questions / Aims

Compared to conventional irrigation regimes, do those promoting dEMCs release during NSRCT in patients diagnosed with apical periodontitis significantly:

i) Improve success-rates of endodontic treatment? ii) Increase bony healing of periradicular lesions? ii) Reduce periradicular pro-inflammatory mediator activity within PTF?

- Methodology

A triple blinded parallel group randomised controlled trial design will be used in accordance with CONSORT guidelines to answer the aforementioned in vivo research question . Sample sizes will be based on other clinical trials which have evaluated periradicular inflammatory mediator activity during NSRCT as no prior data exists for a power calculation. Forty systemically fit adult patients diagnosed with asymptomatic apical periodontitis in single-rooted permanent teeth will be recruited, blinded and block-randomised into control or test groups using an online random number generator with allocation concealment (n=20). Thereafter, they will receive two-visit NSRCT with a standardised irrigant regime that either promotes release of dEMC (17% EDTA solution only) or is considered conventional (5.25% NaOCl solution only). A single operator will provide treatment but be blinded to the intervention alongside patients and assessors. Participants will be reviewed 12 months post-treatment before exiting the trial. All data will be analysed on an intention to treat basis and the following outcome measures/techniques will be used to determine the clinical effectiveness of the test irrigant regime:

i) Treatment success-rates: Clinical and plain-film radiographic information will be collected from participants prior to, immediately after and 12 month post-operatively by a single calibrated operator. Success criteria for NSRCT defined by the European Society of Endodontology Quality Guidelines (i.e. "favourable", "uncertain" and "unfavourable") will then be used to determine if the test irrigant regime results in more favourable treatment outcomes.

ii) Volumetric CBCT image analysis of periradicular bony healing: Pre- and 12 month post-operative CBCT radiographs will be obtained under standardised conditions and uploaded onto InVesalius 3D image-analysis software. A semi-automated threshold algorithm will then be applied to segment the periradicular lesion and calculate its volume (mm3). Pre- and post-operative values will be used to more precisely determine if the test irrigant regime results in significantly greater periradicular bony healing.

ii) Multiplex ELISA array: Exudate will be collected from periradicular tissues via the root canal following endodontic access (baseline), chemo-mechanical preparation, 2-weeks intracanal medication and immediately prior to obturation with an optimised paper-point sampling/eluting protocol. Samples will be analysed with a multiplex ELISA assay, which will determine the concentration of 40 inflammatory analytes known to participate in the pathophysiology of apical periodontitis. Statistical comparisons will determine if the test irrigant regime significantly reduces concentrations of pro-inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with apical periodontitis
* Single rooted permanent teeth
* Medically fit
* Adult patients (≥ 18)
* Voluntarily consent to partake in the study

Exclusion Criteria:

* Teeth in sextants with active periodontal disease (i.e. pocketing of ≤ 5 mm)
* Tooth unable to retain a rubber dam
* Teeth that have had previous endodontic treatment
* Root apex in close proximity to the maxillary sinus
* Patients who have had antimicrobial therapy within 3 months prior to the screening clinic
* Pregnant or breastfeeding women
* Do not have capacity to consent
* Patients that have systemic condition that would reduce immune function

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Treatment Success Rate | 12 months
  Clinical/radiographic information (i.e. absence of pain and resolution of swelling, pain on percussion / palpation and reduction in size of periradicular lesion) will be collected at baseline and again at a 12 month follow-up. Treatment success will be determined based on criteria outlined by the European Society of Endodontology (ESE) Quality Guidelines for NSRCT (2006). In these criteria, outcomes are defined as being "favourable" (absence of pain, swelling and other symptoms, no sinus tract, no loss of function and radiological evidence of a complete healing), "uncertain" (absence of pain, swelling and other symptoms, no sinus tract, no loss of function and radiographic evidence of some healing) and finally "unfavourable" (tooth associated with clinical signs and symptoms of infection such as pain and swelling, sinus tract, loss of function and no radiographic evidence of healing.

SECONDARY OUTCOMES:
Profile of periradicular inflammatory mediators | 14 days
  To analyse inflammatory mediator activity. Periradicular tissue fluid will be retrieved from the peri-radicular tissues through the root canal with a paper point and the concentration of various inflammatory mediators will be quantified via a multiplex bead-based assay technique.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip L Tomson, PhD, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham Dental Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Virdee SS, Bashir N, Camilleri J, Cooper PR, Tomson PL. Exploiting Dentine Matrix Proteins in Cell-Free Approaches for Periradicular Tissue Engineering. Tissue Eng Part B Rev. 2022 Aug;28(4):707-732. doi: 10.1089/ten.TEB.2021.0074. Epub 2021 Oct 7. PMID 34309453